CLINICAL TRIAL: NCT05481047
Title: Arterial Hypotension and Regional Cerebral Oxygen Saturation During Major Abdominal Surgery. A Randomized Controlled Trial
Brief Title: Prevention or Treatment of Arterial Hypotension and Oxygen Cerebral Saturation During Major Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, RUSSO ANDREA, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5079
Record Dates: First submitted 2022-07-22; First posted 2022-08-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hypotension During Surgery; Hemodynamic Instability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prevention (Experimental): investigator will prevent intraoperative arterial hypotension based on HPI index
  Interventions: Device: HPI
- treatment (No Intervention): investigators will treat intraoperative arterial hypotension based on standard hemodynamic parameters

INTERVENTIONS:
Device: HPI — based on HPI values, clinicians will administer drugs or fluids in order to avoid arterial hypotension
  Arms: prevention

SUMMARY:
In this study investigators will explore the association between intraoperative arterial hypotension and cerebral oxygen saturation in patients scheduled for major abdominal surgery. Investigators will assign patients to control or interventional group. In this last group arterial hypotension will be avoided based on a HPI (Hypotension Predictive Index) protocol. In the control group arterial hypotension will be promptly treated according to hemodynamic variables.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for abominal surgery

Exclusion Criteria:

* Emergency surgery
* end-stage renal disease
* pregnancy
* obesity
* atrial fibrillation
* previous cerebral ischaemia
* central nervous system disorders

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Cerebral tissue oximetry | immediately after surgery
  the difference among the two groups of the percentage value of the median value of Cerebral Oxygen Saturation measured by the near-nfrared spectroscopic technology (Foresight sensor)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Russo, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli
Locations (1):
- Fondazione Policlinico Universitairo Agostino Gemelli, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided